CLINICAL TRIAL: NCT03668392
Title: Asparaginase Activity Monitoring (AAM) in Adult Patients With Acute Lymphoblastic Leukemia (ALL)
Acronym: ALL2518
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment rate
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALL2518; 2018-003517-17 (EudraCT Number)
Record Dates: First submitted 2018-09-11; First posted 2018-09-12 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients on Oncospar (Experimental)
  Interventions: Drug: Asparaginase

INTERVENTIONS:
Drug: Asparaginase — Measurement of serum Asparaginase activities during therapy, in terms of intensity and duration, as surrogate parameter for asparaginase depletion.

SUMMARY:
In order to understand how pharmacokinetics and immunological inactivation affect the therapeutic efficacy of Asparaginase (ASP), it is of help and advised in the frame of clinical font-line protocols to monitor the enzymatic activity by measuring the serum ASP levels in the days following the administration of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent according to ICH/EU/GCP and national local laws
* Age 18 - 65 years
* Diagnosis of untreated Ph- ALL entering treatment including PEG-ASP in induction and consolidation
* ECOG performance status 0-2, unless a performance of 3 is unequivocally caused by the disease itself and not by pre-existing comorbidity, and is considered and/or documented to be reversible following the application of antileukemic therapy and appropriate supportive measures

Exclusion Criteria:

* Diagnosis of Burkitt's leukemia
* Down's syndrome
* Adults with Ph+ ALL
* Pre-existing, uncontrolled pathology such as heart failure (congestive/ischemic, acute myocardial infarction within the past 3 months, untreatable arrhythmias, NYHA classes III and IV)
* Severe liver disease with serum bilirubin >3 mg/dL and/or ALT >3 x upper normal limit (unless attributable to ALL)
* Kidney function impairment with serum creatinine >2 mg/dL (unless attributable to ALL)
* Severe neuropsychiatric disorder that impairs the patient's ability to understand and sign the informed consent, or to cope with the intended treatment plan
* Presence of serious, active, uncontrolled infections
* Pre-existing HIV positive serology (i.e. already known before enrolment). If HIV positivity is detected after enrolment, the patient is put off study.
* Pregnancy
* Men and women should use effective contraception during treatment and for at least 6 months after Asparaginase discontinuation. As a precautionary measure, breast-feeding should be discontinued during treatment with Asparaginase and should not be restarted after discontinuation of Asparaginase

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with active serum Asparaginase | After 8 months from study entry

CONTACTS AND LOCATIONS:
Overall Officials: Marco Vignetti, Study Chair — Dipartimento di Biotecnologie Cellulari ed Ematologia - Università degli Studi "Sapienza" di Roma
Locations (7):
- Italy (7):
  - Aou Ospedali Riuniti "Umberto I - G.M. Lancisi - G. Salesi"- Ancona - Sod Clinica Ematologica, Ancona
  - Aso S. Croce E Carle - Cuneo - Sc Ematologia, Cuneo
  - Asl Roma 2, Ospedale S. Eugenio- Ospedale S.Eugenio - Uoc Ematologia, Roma
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia - Università Degli Studi Di Torino, Torino
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia 2, Torino
  - Asui Di Udine - Presidio Ospedaliero "Santa Maria Della Misericordia" - Clinica Ematologica, Udine
  - Aou Integrata Di Verona, Policlinico G.B. Rossi - Uoc Ematologia, Verona

IPD SHARING:
Plan to Share IPD: Undecided